CLINICAL TRIAL: NCT07232680
Title: Integrated Prospective Analysis of Radiomic and Immunologic Signatures in Nasopharyngeal Carcinoma Treated With Proton or Photon Radiotherapy
Brief Title: Prospective Immuno-Radiomic Profiling in Nasopharyngeal Carcinoma Treated With Proton or Photon Chemoradiotherapy
Acronym: IMPRINT
Status: Recruiting | Type: Observational
Sponsor: Cheng-En Hsieh (Other)
Responsible Party: Sponsor-Investigator, Cheng-En Hsieh, Associate Professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: 202501031A3
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: NPC Patients; Nasopharyngeal Cancinoma (NPC)
Keywords: NPC; proton radiotherapy; photon radiotherapy; proton beam therapy; IMPT; IMRT; IMAT; chemoradiation; Immune response; Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples (including plasma and cellular components) will be collected at baseline, 6-8 weeks, and 3-4 months after the initiation of radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Proton chemoradiotherapy: Proton chemoradiotherapy: 69.96 cobalt Gray equivalent (CGE) in 33 fractions
  Interventions: Radiation: Proton chemoradiotherapy
- Photon chemoradiotherapy: Photon chemoradiotherapy: 69.96 Gy in 33 fractions
  Interventions: Radiation: Photon chemoradiotherapy

INTERVENTIONS:
Radiation: Proton chemoradiotherapy — Concurrent chemoradiotherapy will be delivered using intensity modulated proton therapy, with a total dose of 69.96 CGE administered in 33 fractions.
  Groups: Proton chemoradiotherapy
Radiation: Photon chemoradiotherapy — Concurrent chemoradiotherapy will be delivered using photon-based volumetric modulated arc therapy, with a total dose of 69.96 Gy administered in 33 fractions.
  Groups: Photon chemoradiotherapy

SUMMARY:
To prospectively investigate and integrate radiomic and immunologic signatures in patients with nasopharyngeal carcinoma (NPC) treated with either proton or photon radiotherapy, with the aim of identifying biomarkers associated with treatment response, toxicity, and long-term outcomes.

DETAILED DESCRIPTION:
This is a non-randomized, single-center, phase II prospective trial enrolling patients with stage I-III NPC undergoing definitive proton or photon chemoradiotherapy. Participants will be followed for ≥2 years after treatment completion to evaluate clinical outcomes and longitudinal biomarker dynamics, including radiomic and immunologic signatures.

Radiotherapy target delineation was performed according to established consensus guidelines. The gross tumor volume (GTV) included all radiologically visible primary tumors and involved lymph nodes. The clinical target volume receiving 69.96 Gy encompassed the GTV with a 0-5 mm margin and may also include the entire nasopharynx. The clinical target volume receiving 59.4 Gy was optionally delineated at the discretion of the treating physician to encompass regions at high risk for microscopic disease spread, including the nasopharynx, nasal cavity, maxillary sinuses, pterygoid plates, parapharyngeal space, retropharyngeal lymph nodes, clivus, skull base, sphenoid sinus, and bilateral upper cervical lymph nodes. The elective neck volumes, receiving 50-54.12 Gy , encompassed the bilateral cervical lymphatic drainage regions. The detailed contour definitions followed the International Consensus Guidelines on Delineation of Clinical Target Volumes at Different Dose Levels for Nasopharyngeal Carcinoma.

Concurrent Chemotherapy Regimens:

1. Cisplatin Based Regimens

   o Dosage: Cisplatin 100 mg/m² IV on Day 1 every 3 weeks during radiotherapy (total 2-3 cycles); Cisplatin 50 mg/m² IV on Day 1 every 2 weeks during radiotherapy (typically 6-8 weeks); Cisplatin 40 mg/m² IV weekly during radiotherapy (typically 6-7 weeks)
2. Carboplatin-Based Regimens o Dosage: Carboplatin AUC 5-6 IV every 3 weeks

The use of induction chemotherapy is allowed in locally advanced NPC

1. TPF Regimen (Docetaxel + Cisplatin + 5-Fluorouracil)

   * Docetaxel: 75 mg/m² IV on Day 1
   * Cisplatin: 75 mg/m² IV on Day 1
   * 5-FU: 750-1000 mg/m²/day continuous IV infusion on Days 1-5
   * Cycle: Every 3 weeks × 2-3 cycles
2. GP Regimen (Gemcitabine + Cisplatin)

   * Gemcitabine: 1000 mg/m² IV on Days 1 and 8
   * Cisplatin: 80 mg/m² IV on Day 1
   * Cycle: Every 3 weeks × 2-3 cycles
3. TP Regimen (Docetaxel + Cisplatin)

   * Docetaxel: 75 mg/m² IV on Day 1
   * Cisplatin: 75 mg/m² IV on Day 1
   * Cycle: Every 3 weeks × 2-3 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent.
2. Pathologically confirmed diagnosis of nasopharyngeal carcinoma
3. Age ≥18 years
4. ECOG performance status 0-1
5. Patients with AJCC v.9 stage I-III disease who undergo chemoradiotherapy
6. Adequate bone marrow, liver, and renal function within 4 weeks before study registration

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 2.5 mg/dL
   * Serum albumin >2.8 g/dL
   * Serum creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

1. Presence of distant metastasis
2. Patients with AJCC v.9 cT1N0M0 disease who undergo radiotherapy alone.
3. Synchronous or prior invasive malignancy, unless disease-free for at least 2 years.
4. Prior radiotherapy to the head and neck region
5. Presence of severe major organ dysfunction
6. Pregnant women or women of childbearing potential who are unwilling to use medically acceptable contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AJCC 9th edition stage I-III nasopharyngeal carcinoma undergoing definitive chemoradiotherapy using either proton or photon radiotherapy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2031-08-15 (Estimated); Study Completion 2034-08-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival is defined as the time from signing the informed consent to death from any cause.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Progression free survival is defined as the time from signing the informed consent to the first occurrence of disease progression or death from any cause (whichever occurs first) according to RECIST1.1
Time to progression | 2 years
  Time to progression is defined as the time from signing the informed consent to the first occurrence of disease progression according to RECIST1.1.
Incidence and severity of adverse events | 5 years
  Acute and late adverse events will be graded using CTCAE v5

OTHER OUTCOMES:
Changes of myeloid-derived suppressor cell levels | 4 months
  The levels of myeloid-derived suppressor cells (MDSCs) in peripheral blood will be analyzed at baseline, 6-8 weeks, and 3-4 months following the initiation of radiotherapy.
Changes in MRI radiomic parameters | 4 months
  Radiomic features will be extracted from MRI obtained pre-treatment and at 3-4 months post-chemoradiotherapy; feature changes will be computed as absolute (Δf = fpost - fpre) and percent change (Δ% = 100 × (fpost - fpre) / fpre)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Cheng En Hsieh, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The sharing of individual participant data (IPD) will be conducted only after obtaining approval from the Institutional Review Board (IRB) and in accordance with applicable ethical and data protection regulations.